CLINICAL TRIAL: NCT05349903
Title: Impact of Slowly Digestible Carbohydrates on the Gut-brain Axis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Collaborators: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Principal Investigator, Bruce R. Hamaker, Distinguished Professor of Food Science, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB-2020-986
Record Dates: First submitted 2021-10-06; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Appetitive Behavior; Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Appetitive Behavior; Obesity; Diabetes Mellitus, Type 2 | interventions — Flour; Inulin; epigallocatechin gallate

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Rice flour (Experimental): Rapidly digestible control
  Interventions: Other: Rice flour
- Alternanoligosaccharide 15 (Experimental)
  Interventions: Other: Alternanoligosaccharide 15
- Waxy potato starch (Experimental)
  Interventions: Other: Waxy potato starch
- Combination of waxy potato starch and epigallocatechin gallate (EGCG) (Experimental)
  Interventions: Other: Waxy potato starch + epigallocatechin gallate (EGCG)
- Combination of chickpea flour and epigallocatechin gallate (EGCG) (Experimental)
  Interventions: Other: Chickpea flour + epigallocatechin gallate (EGCG)
- Inulin (Experimental)
  Interventions: Other: Inulin

INTERVENTIONS:
Other: Rice flour — Rice flour made into rice porridge will be tested for postprandial glycemic response, gut hormone levels, gastric emptying rate, appetitive response, and fermentability.
  Arms: Rice flour
Other: Alternanoligosaccharide 15 — Alternanoligosaccharide 15 incorporated into rice porridge will be tested for postprandial glycemic response, gut hormone levels, gastric emptying rate, appetitive response, and fermentability.
  Arms: Alternanoligosaccharide 15
Other: Inulin — Inulin incorporated into rice porridge will be tested for postprandial glycemic response, gut hormone levels, gastric emptying rate, appetitive response, and fermentability.
  Arms: Inulin
Other: Waxy potato starch — Retrograded waxy potato starch made into porridge meal will be tested for postprandial glycemic response, gut hormone levels, gastric emptying rate, appetitive response, and fermentability.
  Arms: Waxy potato starch
Other: Waxy potato starch + epigallocatechin gallate (EGCG) — A combination of retrograded waxy potato starch and EGCG made into porridge meal will be tested for postprandial glycemic response, gut hormone levels, gastric emptying rate, appetitive response, and fermentability.
  Arms: Combination of waxy potato starch and epigallocatechin gallate (EGCG)
Other: Chickpea flour + epigallocatechin gallate (EGCG) — A combination of chickpea flour and EGCG made into porridge meal will be tested for postprandial glycemic response, gut hormone levels, gastric emptying rate, appetitive response, and fermentability.
  Arms: Combination of chickpea flour and epigallocatechin gallate (EGCG)

SUMMARY:
Our laboratory is investigating the physiological outcomes and health benefits of the consumption of high-quality carbohydrates. One important aspect of the high-quality carbohydrate characteristics is a slow and sustained digestion and glucose release to the blood. In the proposed study, the investigators will evaluate the consumption of different types of slowly digestible carbohydrates (SDCs) and their beneficial effects including moderation of the glycemic response profile (postprandial glycemic response, PPGR) and stimulation of the gut-brain axis, which controls appetite and food intake. This stimulation will be evaluated in terms of second-meal food intake and the circulatory level of appetite-suppressing gut hormones (such as glucagon-like peptide-1).

ELIGIBILITY:
Inclusion Criteria:

* BMI 18.5 - 25 kg/m2
* Stable weight for the past 3 months (i.e. +/- 2..5 kg)

Exclusion Criteria:

* Pregnant or nursing women
* Diabetic
* Individuals with history of gastrointestinal disease

Ages: 22 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-10 (Actual); Primary Completion 2022-02-24 (Actual); Study Completion 2022-02-24 (Actual)

PRIMARY OUTCOMES:
Postprandial glycemic response | Acute study: [4 hours of measurement after consumption of test food]
  Blood plasma glucose will be measured, (AUC)
Postprandial glycemic response | Acute study: [4 hours of measurement after consumption of test food]
  Blood plasma glucose will be measured, (C max)
Postprandial glycemic response | Acute study: [4 hours of measurement after consumption of test food]
  Blood plasma glucose will be measured, (t max)
Postprandial plasma gut hormone response | Acute study: [4 hours of measurement after consumption of test food]
  Blood plasma glucagon-like peptide-1 and insulin will be measured, (AUC)
Postprandial plasma gut hormone response | Acute study: [4 hours of measurement after consumption of test food]
  Blood plasma glucagon-like peptide-1 and insulin will be measured, (C max)
Postprandial plasma gut hormone response | Acute study: [4 hours of measurement after consumption of test food]
  Blood plasma glucagon-like peptide-1 and insulin will be measured, (t max)

SECONDARY OUTCOMES:
Gastric emptying rate | Acute study: 4 hours of measurement after consumption of test food]
  Breath test will be performed using 13C-acetate mixed into test meals
Appetite ratings (Visual Analog Scale, VAS) | Acute study: [4 hours of measurement after consumption of test food]
  Hunger and fullness scores will be measured using a 10-cm scale (0 = weakest feeling of hunger or fullness and 10 = strongest feeling of hunger or fullness) after consumption of test food. Weaker feelings of hunger and stronger feelings of fullness indicate better outcomes.
Food Intake of the next meal | Acute study: After the consumption a second meal [4 hours later after consuming the first meal]
  At the end of the 4 hour window, participants will be given a large second meal for consumption and the amount of consumed food (food intake) will be estimated.
Breath hydrogen (fermentability) | Acute study: [4 hours of measurement after consumption of test food]
  Breath samples will be collected in 15-minute intervals for 4 hours after consumption of test food and analyzed for hydrogen levels using a breath analyzer. Breath hydrogen levels are indicative of a food's fermentability.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce R Hamaker, PhD, Principal Investigator — Purdue University
Locations (1):
- Purdue University, West Lafayette, Indiana, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to other researchers.